CLINICAL TRIAL: NCT01641575
Title: A Phase I Open-Label, Ascending Dose Cohort Study of Gemcitabine Elaidate and Cisplatin in Patients With Advanced Solid Tumors Followed by an Expanded Cohort of Patients With Stage IIIb/IV NSCLC.
Brief Title: A Dose Ascending Study of Gemcitabine Elaidate (CO-101) in Combination With Cisplatin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Registrational study did not meet endpoint so entire program (including CO-101-011) was terminated.
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-101-011
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Solid Tumor; Non-small-cell Lung Cancer; Lung Cancer
Keywords: CO-1.01; CO-101; gemcitabine elaidate; hENT1; nucleoside equilibrative transporter; solid tumor; non-small-cell lung cancer; NSCLC; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; CP 4126

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CO-1.01 and Cisplatin (Experimental)
  Interventions: Drug: CO-1.01 and Cisplatin

INTERVENTIONS:
Drug: CO-1.01 and Cisplatin — CO-1.01 administered over 30 minutes followed by 75 mg/ml Cisplatin over 2 hours (both intravenous) on C1D1. CO-1.01 administered intravenously over 30 minutes on C1D8.
  Other Names: Gemcitabine elaidate

SUMMARY:
The purpose of the first part of the study is to evaluate the safety, tolerability, and pharmacokinetics of ascending doses of gemcitabine elaidate in combination with cisplatin given to patients with advanced solid tumors, and to select a dose for further evaluation in the second part of the study.

The purpose of the second part of the study is to determine the safety, tolerability, and exploratory clinical activity of gemcitabine elaidate in combination with cisplatin given to patients with Stage IIIb/IV non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The chemotherapy doublet of cisplatin and gemcitabine is an effective regimen for solid tumors including NSCLC. Entry of gemcitabine into tumor cells has been shown to be dependent on specific membrane transporter proteins, particularly human equilibrative nucleoside transporter 1 (hENT1). Patients with low tumor hENT-1 expression may respond poorly to gemcitabine-containing chemotherapy. Gemcitabine elaidate (CO-1.01) is a fatty acid derivative of gemcitabine, and can enter cells in the absence of hENT1. CO-1.01 therefore, may overcome hENT1-mediated resistance to gemcitabine.

CO-1.01 is currently being evaluated as a single agent in a pivotal randomized trial in 360 patients with metastatic pancreatic adenocarcinoma. The appropriate dose of CO-1.01 when given as part of combination therapy with a platinum agent such as cisplatin is not yet known. The objectives of this study are to:

* determine the maximum tolerated dose (MTD) of CO-1.01 when combined with a fixed dose of cisplatin in patients with solid tumors
* select a recommended dose (RD) for dose expansion in patients with Stage IIIb/IV NSCLC
* explore clinical activity of CO-1.01 in patients with Stage IIIb/IV NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign institutional review board/independent ethics committee-approved informed consent form (ICF) prior to any study-specific evaluation
* Life expectancy of at least 3 months
* ECOG performance status of 0 to 1
* ≥ 18 years at the time ICF is signed
* Adequate hematological and biological function
* Histologically or cytologically confirmed solid tumor malignancy (Part 1 only)
* Histologically or cytologically confirmed stage IIIb/IV NSCLC (Part 2 only)

Exclusion Criteria:

* Symptomatic central nervous system metastases
* Concomitant treatment with prohibited medications, e.g. other chemotherapy, radiation, hormonal treatment (excepting corticosteroids), or immunotherapy ≤ 14 days prior to CO-1.01 treatment
* Treatment with a previous regimen of CO-1.01
* Participation in another therapeutic clinical study within 14 days of enrollment or during this clinical study
* Surgical procedures ≤ 14 days prior to CO-1.01 administration
* History of allergy to gemcitabine, gemcitabine elaidate or eggs
* Known allergic/hypersensitivity reaction to cisplatin, other platinum agent, or platinum containing compounds
* Peripheral neuropathy ≥ Grade 1
* Females who are pregnant or breastfeeding
* Refusal to use adequate contraception for fertile patients
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
* Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT)(Part 1) | From time taking first dose of CO-1.01 (Cycle 1 Day 1) through last day of Cycle 1 (Cycle 1 Day 21), an expected average of 6 weeks.
Adverse events (Description of event in medical terminology, Intensity, Relationship to drug, Outcome, and/or Follow up )(Part 2) | From time of signing informed consent form through 28 days after last dose of CO-1.01, an expected average of 7 weeks
Clinical Laboratory Abnormalities (ANC, Platelets, Hemoglobin, AST/ALT, Bilirubin, Creatinine clearance)(Part 2) | For Cycle 1: Day 1, Day 8, Day 15. For subsequent cycles: Day 1, Day 8.
ECG Abnormalities (Part 2) | Screening (within 2 weeks of Cycle 1 Day 1)

SECONDARY OUTCOMES:
PK parameters for CO-1.01 and its metabolites in plasma and urine (AUC, Cmax, Tmax, half life, kel, Vss, Cl, and MRT) (Part 1) | Cycle 1: Day 1, Day 8
Adverse events (Description of event in medical terminology, Intensity, Relationship to drug, Outcome, and/or Follow up )( (Part 1) | From time of signing informed consent form through 28 days after last dose of CO-1.01, an expected average of 7 weeks
Clinical Laboratory Abnormalities (ANC, Platelets, Hemoglobin, AST/ALT, Bilirubin, Creatinine clearance)(Part 1) | For Cycle 1: Day 1, Day 8, Day 15. For subsequent cycles: Day 1, Day 8.
ECG abnormalities (Part 1) | Screening (within 2 weeks of Cycle 1 Day 1)
Overall response rate (ORR)(Part 2) | Screening (within 2 weeks of Cycle 1 Day 1); prior to start of cycles 3,5,7; every 3 cycles thereafter
Duration of response (Part 2) | Screening (within 2 weeks of Cycle 1 Day 1); prior to start of cycles 3,5,7; every 3 cycles thereafter
Progression-free survival (PFS)(Part 2) | Screening (within 2 weeks of Cycle 1 Day 1); prior to start of cycles 3,5,7; every 3 cycles thereafter
Tumor hENT1 expression (Part 2) | Screening (within 2 weeks of Cycle 1 Day 1)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Florida Cancer Specialists, Sarasota, Florida
  - Tennessee Oncology, Nashville, Tennessee
- United Kingdom (2):
  - University College London Cancer Institute, London, London
  - The Beatson West, Glasgow, Scotland